CLINICAL TRIAL: NCT02641834
Title: Prevention of Cardiovascular Disease With the Vegetarian Diet: the CARDIVEG Study
Brief Title: Prevention of Cardiovascular Disease With Med or Veg Diets
Acronym: CARDIVEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Associate Professor of Clinical Nutrition, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CAR-123-VEG
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Results first posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Disease
Keywords: diet; vegetarian; cardiovascular risk
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Diet, Vegetarian; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Veg Group (Experimental): Group that starts with the Vegetarian diet
  Interventions: Other: Vegetarian diet; Other: Mediterranean diet
- Med group (Active Comparator): Group that starts with the Mediterranean diet
  Interventions: Other: Vegetarian diet; Other: Mediterranean diet

INTERVENTIONS:
Other: Vegetarian diet — 7-days dietary profile with an isocaloric Vegetarian diet for 3 months
Other: Mediterranean diet — 7-days dietary profile with an isocaloric Mediterranean diet for 3 months

SUMMARY:
The study is a randomized, open, cross-over trial designed to test whether a vegetarian diet would benefit the cardiovascular risk profile of the participants, compared with a Mediterranean diet.

DETAILED DESCRIPTION:
Nutrition is able to substantially alter the health status of the general population. In industrialized countries such as Italy the most important association between diet and health is certainly the relationship with cardiovascular disease, the leading cause of death and disability. The ability to identify with certainty, therefore, the relationship between diet and cardiovascular disease appears to be a key element in the implementation of specific primary prevention strategies.

Cardiovascular diseases would be the result of interactions between genetics and environmental factors. Many studies have evaluated the associations between food groups, foods, or nutrients and chronic diseases, and a consensus about the role of nutritional factors in the etiology of common diseases, such as cardiovascular and neoplastic diseases, has gradually emerged. Recent studies have been focused on examining the impact of a whole dietary approach rather than on isolating single nutrients; it is recognized that analyses of single nutrients ignore the important and complex interactions between components of a diet and, more importantly, because people do not eat isolated nutrients.

The optimal dietary strategy for the prevention of chronic degenerative diseases remains a challenging and a highly relevant preventive health issue. Over the last years, numerous evidence on the existing relationship between nutrition and chronic degenerative diseases have led investigators to search for the optimal dietary pattern to maintain a good health status. Several models of diet have been imposed on public attention, but those that got the most interest are certainly Mediterranean and vegetarian diets. These dietary patterns seem to exert protective effects on blood pressure, lipid profiles, cardiovascular diseases and metabolic parameters.

The term Mediterranean diet has been widely used to describe the traditional dietary habits of people in Crete, South Italy, and other Mediterranean countries during the decade of the 1960s. Since the first data from the Seven Countries Study, several studies in different populations have established a beneficial role for the main components of the Mediterranean diet on the occurrence of cardiovascular diseases and chronic degenerative diseases. This dietary pattern is characterized by plentiful plant foods (fruits, vegetables, breads, other forms of cereals, beans, nuts, and seeds), olive oil as the principal source of fat, moderate amounts of dairy products (mainly cheese and yogurt), low to moderate amounts of fish and poultry, red meat in low amounts and wine consumed in low to moderate quantities, usually with meals.

The vegetarian diet is a diet that excludes the use of animal foods (meat, fish) in its fresh, preserved and/or processed. The increase in the number of vegetarians is attributable to health, ethical, environmental, and social concerns.

Recently, meta-analysis conducted by our group have revealed, in a population of over than 2 million of people, that a strict adherence to a Mediterranean dietary pattern is associated with a significant improvement in health status, as seen by a significant reduction in overall mortality (10%) and incidence and/or mortality from cardiovascular diseases (9%).

During the past few decades, there has been a gradual abandonment of this dietary pattern by the inhabitants of the Mediterranean basin, especially by the younger generations. Several factors have contributed to this nutrition transition, such as the enhanced commercial availability of food, the urbanization of life, and the overall improvement in socioeconomic conditions in Europe, which has increased the food and energy supply and made food (especially of animal origin) more affordable. Consumption of milk, meat and animal fat products increased in all Mediterranean countries. Moreover, a stressful lifestyle, less time spent on cooking, and the enhanced variety and availability of household appliances have also been proposed as determinants of nutrition transition.

Because of the growing evidence in favor of link between red and processed meat and cardiovascular disease risk, cancer and diabetes, the interest towards vegetarian diets has increased. In the last years, the number of subjects who began to adopt a vegetarian dietary pattern has enormously increased with respect to the past, when the population of vegetarians was limited only to few and selected cohorts. Such increase has been mainly attributed to the supposed beneficial effect of this dietary pattern versus the occurrence of diseases.

Health benefits of Mediterranean and vegetarian diets have been widely described in case-control and prospective cohort studies during the last 50 years. There are several beneficial nutrients that are abundant in these diets, such as monounsaturated fatty acids, high amounts of fiber and antioxidants and low intake of total and saturated fats. However, it is unclear whether established health benefits for vegetarians are attributable to the absence of meat in the diet, the increased consumption of particular food component(s) the pattern of foods eaten within the vegetarian diet or other healthy lifestyle components often associated with vegetarianism.

In a recent systematic review with meta-analysis carried out on over than 130,000 vegetarians, plant-based diet was associated with many health benefits. Main findings were that vegetarian diet determines, among case-control studies, lower levels of the most important risk factor for chronic disease, along with a reduced risk of occurrence for ischemic heart disease (-25%) when cohort prospective studies were taken into account.

Currently there are no randomized controlled trials to compare, in a high-risk group of patients with risk factors for cardiovascular disease, the efficacy of nutritional interventions based on Mediterranean and vegetarian dietary patterns. From this comparison it would may be possible to obtain interesting results in order to identify the optimal diet for prevention of cardiovascular diseases.

OBJECTIVES:

The primary aim of the study is to compare the effects of vegetarian diet on risk markers (anthropometric and biochemical measures) associated with cardio-metabolic diseases (CMD) after a 3-month dietary-intervention phase, compared with a Mediterranean diet.

Secondary objectives of the study are:

* To improve knowledge about the pathophysiological role of vegetarian and Mediterranean diets in cardiovascular prevention
* To evaluate the feasibility and degree of adherence to a dietary substitution with vegetarian diet in a omnivorous population
* To evaluate the ability of a nutrition education intervention to reduce fresh and processed meat consumption in subjects at high cardiovascular risk, in order to enhance health and quality of life
* To explore the impact of food prices on consumption and to evaluate the overall cost of buying food products in different dietary patterns

STUDY DESIGN The study is a randomized, open, cross-over trial designed to test whether a vegetarian diet would benefit the cardiovascular risk profile of the participants, compared with a Mediterranean diet.

The eligible participants are randomly divided into two groups, each assigned to either the experimental group (Group 1), which receives a vegetarian diet, or the control group (Group 2), which receives a Mediterranean diet. Following the first intervention phase, the subjects are crossed over in order to obtain the second intervention phase. Both diets are isocaloric and lasting three months each. The whole trial includes five clinical visits.

STUDY POPULATION Subjects in primary prevention with low-middle cardiovascular risk (1-5% according to the guidelines of the European Society of Cardiology), determined by the presence of BMI >o=25 kg/m2 and no more than other 2 concomitant metabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Willing and able to give informed consent
3. Presence of at least one of the following risk factors for cardiovascular disease (European Society of Cardiology guidelines on cardiovascular disease prevention):

   * BMI >o= 25 kg/m2
   * Waist circumference > 88 cm (women) or > 102 cm (men)
   * Circulating levels of total cholesterol > 190 mg/dL, non-drug treatment (measured no more than 3 months prior to the start of the study)
   * Circulating levels of LDL cholesterol > 115 mg/dL, non-drug treatment (measured no more than 3 months prior to the start of the study)
   * Levels of circulating triglycerides > 150 mg/dL, non-drug treatment (measured no more than 3 months prior to the start of the study)
   * Circulating levels of fasting blood glucose > 110 and < 126 mg/dL, non-drug treatment (measured no more than 3 months prior to the start of the study)
4. Wiling to participate in a randomized study comparing two dietary profiles, one of which is a vegetarian dietary pattern
5. Successfully completed 3-day food diary
6. Wiling to be contacted at least twice during the study period to evaluate diet compliance
7. Wiling to provide blood and fecal samples

Exclusion Criteria:

1. Presence of current serious illness or unstable condition that requires physician supervision of diet or physical activity (e.g., recent myocardial infarction, chronic liver disease, inflammatory bowel diseases)
2. Pregnancy or intention to become pregnant in next 18 months
3. Lactation
4. Current or recent (past 6 months) participation in weight loss treatment program or use of weight loss medication
5. Reporting no regular intake of meat, fish, or poultry for past month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Casini, MD, Study Director — Unit of Clinical Nutrition, University Hospital of Careggi
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pagliai G, Tristan Asensi M, Dinu M, Cesari F, Bertelli A, Gori AM, Giusti B, Marcucci R, Sofi F, Colombini B. Effects of a dietary intervention with lacto-ovo-vegetarian and Mediterranean diets on apolipoproteins and inflammatory cytokines: results from the CARDIVEG study. Nutr Metab (Lond). 2024 Feb 1;21(1):9. doi: 10.1186/s12986-023-00773-w. PMID 38302995
- [Derived] Ronca A, Pellegrini N, Pagliai G, Dinu M, Manfredini M, Incerti M, Favari E, Sofi F. Effects of a dietary intervention with Mediterranean vs lacto-ovo vegetarian diets on HDL function: Results from the CARDIVEG study. Nutr Metab Cardiovasc Dis. 2023 Mar;33(3):651-658. doi: 10.1016/j.numecd.2022.11.012. Epub 2022 Nov 24. PMID 36642608
- [Derived] Sofi F, Dinu M, Pagliai G, Cesari F, Gori AM, Sereni A, Becatti M, Fiorillo C, Marcucci R, Casini A. Low-Calorie Vegetarian Versus Mediterranean Diets for Reducing Body Weight and Improving Cardiovascular Risk Profile: CARDIVEG Study (Cardiovascular Prevention With Vegetarian Diet). Circulation. 2018 Mar 13;137(11):1103-1113. doi: 10.1161/CIRCULATIONAHA.117.030088. Epub 2018 Feb 26. PMID 29483085
- [Derived] Sofi F, Dinu M, Pagliai G, Cesari F, Marcucci R, Casini A. Mediterranean versus vegetarian diet for cardiovascular disease prevention (the CARDIVEG study): study protocol for a randomized controlled trial. Trials. 2016 May 4;17(1):233. doi: 10.1186/s13063-016-1353-x. PMID 27145958

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Veg Group | Med Group
Started | 60 | 58
Completed | 50 | 50
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veg Group | Med Group | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 9 | 7 | 16
Age, Continuous [Median (Full Range); unit: years] | 49.5 [24 to 70] | 52 [21 to 75] | 50 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 43 | 92
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  Italy | 60 | 58 | 118

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Weight From Baseline
Description: Changes in Body Weight From Baseline
Time Frame: baseline and 6 months
Population: All data were treated as paired samples from a crossover study. The 2 interventions were analyzed combining the results obtained in the 2 phases of both groups. As a total of 107 participants completed ≥1 phase of intervention and were included in the analysis, the overall number of participants in each dietary group is greater than the number stated in the participant flow.
Measure: Geometric Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
Kilograms | -1.88 [-2.42 to -1.35] | -1.77 [-2.29 to -1.25]

2. Secondary Outcome: Changes in Fat Mass From Baseline
Description: Changes in fat mass from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of fat mass
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
percentage of fat mass | -1.23 [-1.67 to -0.80] | -1.46 [-1.93 to -1.01]

3. Secondary Outcome: Changes in BMI From Baseline
Description: Changes in BMI from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
kg/m^2 | -0.64 [-0.84 to -0.43] | -0.67 [-0.86 to -0.47]

4. Secondary Outcome: Changes in Total Cholesterol From Baseline
Description: Changes in total cholesterol from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
mg/dL | -5.34 [-10.24 to -0.73] | -0.11 [-4.36 to 4.09]

5. Secondary Outcome: Changes in LDL Cholesterol From Baseline
Description: Changes in LDL cholesterol from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
mg/dL | -6.98 [-11.06 to 2.16] | 2.12 [-2.26 to 5.60]

6. Secondary Outcome: Changes in Triglycerides From Baseline
Description: Changes in triglycerides from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
mg/dL | 5.92 [-1.16 to 16.41] | -6.78 [-14.76 to -2.72]

7. Secondary Outcome: Changes in Glucose From Baseline
Description: Changes in glucose from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
mg/dL | 0.54 [-0.97 to 2.43] | 0.27 [-1.13 to 1.53]

8. Secondary Outcome: Changes in TBARS From Baseline
Description: Changes in TBARS from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
pg/mL | -0.39 [-0.65 to -0.09] | -0.32 [-0.65 to -0.09]

9. Secondary Outcome: Changes in L-derived ROS From Baseline
Description: Changes in L-derived ROS from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: RFU
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
RFU | -59.62 [-105.17 to 6.72] | -17.56 [-79.89 to 26.32]

10. Secondary Outcome: Changes in Interleukin-17 From Baseline
Description: Changes in Interleukin-17 from baseline
Time Frame: baseline and 6 months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Veg Group | Med Group
Number analyzed (Participants) | 104 | 103
pg/mL | 1.39 [-0.62 to 1.84] | -2 [-3.51 to -0.01]

ADVERSE EVENTS:
Arm/Group | Veg Group | Med Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58

LIMITATIONS AND CAVEATS:
Some limitations are present, such as the limited duration of the study. Studies with a larger population and a longer duration are needed to confirm these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No